CLINICAL TRIAL: NCT02580019
Title: Cell Therapy by Intravenous Injection of Umbilical Cord Derived Mesenchymal Stem Cells After Stroke
Brief Title: Umbilical Cord Derived Mesenchymal Stem Cells Treatment in Ischemic Stroke
Acronym: Recruiting
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hospital307
Record Dates: First submitted 2015-07-02; First posted 2015-10-20 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-07

CONDITIONS: Stroke
Keywords: Cellular therapy; Stroke; Neuronal Plasticity; Recovery; umbilical cord mesenchymal stem cells; Transplantation; Cardiovascular Diseases; Ischemia; Brain Infarction; Brain Ischemia; Cerebrovascular Disorders
MeSH Terms: conditions — Stroke; Cardiovascular Diseases; Ischemia; Brain Infarction; Brain Ischemia; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional stroke treatment (No Intervention): Control group without intervention, whereas they receive conventional stroke treatment that including rehabilitation
- hUC-MSC treatment (Experimental): Patients will receive human umbilical cord mesenchymal stem cells transplantation accompanied with conventional treatment including rehabilitation
  Interventions: Biological: Human umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: Human umbilical cord mesenchymal stem cells — A single dose of 2×107 hUC-MSC will treated to patients, IV, Repeat every weeks for four times.
  Arms: hUC-MSC treatment

SUMMARY:
The study aims at estimating the safety and efficacy of the intravenous injection of human umbilical cord mesenchymal stem cell(hUC-MSC) for patients suffering from ischemic stroke in recent 3 months.

DETAILED DESCRIPTION:
Given the attention paid in recent times, in China and elsewhere, to stroke, which is the leading cause of acquired adult disability and has negative effects on patients' quality of life.Therefore,It's little wonder there's much focus there days on treatment of stroke. For the patients who have suffered from ischemic stroke in 3 months, indeed, they have the opportunity to get symptomatic improvement through receiving conventional stroke treatments that including rehabilitation. At the same time, these treatments are ineffective in some cases. Alternatively, the phenomenon of increasing brain plasticity after stroke provoke an essential therapy. Human umbilical cord mesenchymal stem cells treatment enhances a functional improvement after cerebral ischemia, likewise, treament in rodent models are proved effective. Human umbilical cord mesenchymal stem cells therapy performs a role as take the place destroyed cerebral tissue with a stem cells graft. The totality of evidence from trials running umbilical cord mesenchymal stem cells transplanted into patients suffering from ischemic stroke support the safety of this approach. In terms of efficacy, positive results are reported in the majority of the trials.

Our research project involves a development of cell therapy in a phase IIa clinical trial of safety and efficacy in patients (randomised, controlled, open, with 2 parallel groups).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of intracerebral ischemic stroke in three months by Magnetic Resonance Imaging(MRI)
* Patients have received proper treatment within two weeks from the onset of stroke symptoms.
* Age between 18 to 70 years old for men or women
* Patients with persistent neurological deficit .
* Obtaining informed consent signed (after being informed of the purpose, procedure, and venture of this study, the patient or guardian or legal representative must signing the informed consent document for engagement of participation.
* Patients basic situation are allowable to be involved in the program.

Exclusion Criteria:

* Patients with serious extensive stroke, who are unwilling to the risk.
* Patients with serious persistent neurological deficit (NIHSS > 24).
* Medical history of neurological pathology with a deficit as consequence (Rankin < 3 before stroke).
* Patients with serious psychological disease.
* Patients with myocardial infarction in recent 3 months.
* Patients with recurring thromboembolic disease in recentin recent 3 months.
* Patients with organ transplantation.
* Patients with infection history including Human Immunodeficiency Virus(HIV),Human T-cell Leukemia Virus(HTLV), Hepatitis B Virus(HBV), Hepatitis C Virus(HCV),ect.
* Patients receive current immunosuppressive/immunomodulating treatment.
* Patients basic situation are unallowable to be involved in the program.
* Patients who refuse to participate.
* Patients who are inability or unwillingness of individual or legal guardian/representative to give written informed consent.
* Patients who are pregnant or feeding women.
* Patients who are Participating in another therapeutic clinical trial or in period of exclusion of a therapeutic clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of treatment related-adverse events during the study period. | 180 days after transfusion

SECONDARY OUTCOMES:
Comparison of National Institutes of Health stroke scale (NIHSS). | 180 days after the cell treatment.
Comparison of modified Rankin scale (mRS). | 180 days after the cell treatment.
Distinguish of EuroQol 5d (EQ-5D) between pre- and post-treatment 180 days. | 180 days after the cell treatment.
Comparison of infarct size measured by brain MRI. | 180 days after the cell treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Duan Lian, P.H.D, Principal Investigator — Director and Professor, Department of Neurosurgery, Affiliated Hospital(307 Hospital), Academy of Military Medical Science, Beijing, China
Locations (1):
- Department of Neurosurgery,Affiliated Hospital of Academy of Military Medical Sciences(307 Hospital), Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Cheng Q, Zhang Z, Zhang S, Yang H, Zhang X, Pan J, Weng L, Sha D, Zhu M, Hu X, Xu Y. Human umbilical cord mesenchymal stem cells protect against ischemic brain injury in mouse by regulating peripheral immunoinflammation. Brain Res. 2015 Jan 12;1594:293-304. doi: 10.1016/j.brainres.2014.10.065. Epub 2014 Nov 6. PMID 25449888
- [Background] Tsuji M, Taguchi A, Ohshima M, Kasahara Y, Sato Y, Tsuda H, Otani K, Yamahara K, Ihara M, Harada-Shiba M, Ikeda T, Matsuyama T. Effects of intravenous administration of umbilical cord blood CD34(+) cells in a mouse model of neonatal stroke. Neuroscience. 2014 Mar 28;263:148-58. doi: 10.1016/j.neuroscience.2014.01.018. Epub 2014 Jan 18. PMID 24444827
- [Background] Verina T, Fatemi A, Johnston MV, Comi AM. Pluripotent possibilities: human umbilical cord blood cell treatment after neonatal brain injury. Pediatr Neurol. 2013 May;48(5):346-54. doi: 10.1016/j.pediatrneurol.2012.10.010. PMID 23583051
- [Result] Yalvac ME, Rizvanov AA, Kilic E, Sahin F, Mukhamedyarov MA, Islamov RR, Palotas A. Potential role of dental stem cells in the cellular therapy of cerebral ischemia. Curr Pharm Des. 2009;15(33):3908-16. doi: 10.2174/138161209789649439. PMID 19938343
- See also: This review article provides an update role of hUC-MSCs implantation in the treatment of ischemic stroke. — http://journal.hep.com.cn/fmd/EN/Y2015/V9/I1/20
- See also: Human umbilical cord blood-derived mesenchymal stem cell transplantation attenuates severe brain injury by permanent middle cerebral artery occlusion in newborn rats — http://www.nature.com/pr/journal/v72/n3/full/pr201271a.html